CLINICAL TRIAL: NCT05622903
Title: Effect of Cash Benefits on Health Care Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Brigham and Women's Hospital (Other); Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, Sumit Agarwal, Instructor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P000093
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in the treatment group received up to $400 per month.
  Interventions: Other: Cash Benefit
- Control Group (Active Comparator): Participants in the control group did not receive monthly cash benefits.
  Interventions: Other: No Cash Benefit

INTERVENTIONS:
Other: Cash Benefit — Spending from the cards was not restricted to food but could be spent on anything and anywhere Visa was accepted. The debit cards were credited with the first payment on November 18th, 2020 and the second payment on December 18th, 2020. The program continued with monthly credits through August 2021.
  Other Names: Basic Income; Debit Card
  Arms: Treatment Group
Other: No Cash Benefit — No monthly cash benefit.
  Arms: Control Group

SUMMARY:
Using data from the Chelsea Eats program, we propose to study a randomized controlled trial in which the City of Chelsea, Massachusetts held a lottery to allocate cash benefits to its residents for ten months during the first two years of the COVID-19 pandemic. We will analyze the impact of the cash benefit on health care utilization and health.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Chelsea, Massachusetts
* Household income at or below 30% of the U.S. Department of Housing and Urban Development's Area Median Income

Exclusion Criteria:

* See inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3615 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Emergency department use | 10 months
  Count of visits to the emergency department (ED) using the electronic health record

SECONDARY OUTCOMES:
Behavioral health-related ED visit | 10 months
  Visits to the ED with a behavioral health-related diagnosis code
Substance use disorder-related ED visit | 10 months
  Visits to the ED with a substance use disorder-related diagnosis code
Potentially avoidable ED visit | 10 months
  Visits to the ED that are potentially avoidable, categorized as avoidable according to the previously validated New York University algorithm
ED visit resulting in admission to the hospital | 10 months
  Visits to the ED that result in a hospitalization
Outpatient service use | 10 months
  Office visits and visits for other types of outpatient care such as imaging and procedures
COVID vaccination | 10 months
  Binary variable for having received at least one dose of any COVID vaccine by the end of the trial period
Hemoglobin A1c | 10 months
  Continuous measure of diabetes, using the latest available reading or result during trial period
Blood pressure | 10 months
  Continuous measure of blood pressure, using the latest available reading or result during trial period
Weight | 10 months
  Continuous measure of weight, using the latest available reading or result during trial period
Cholesterol | 10 months
  Continuous measure of cholesterol, using the latest available reading or result during trial period

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Agarwal, MD, MPH, Principal Investigator — Brigham and Women's Hospital and Harvard Medical School
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT05622903/Prot_SAP_000.pdf